CLINICAL TRIAL: NCT02760303
Title: Reducing Stress in Adolescents and Young Adults With T1D to Improve Diabetes Care
Brief Title: Reducing Stress in Adolescents and Young Adults With Type 1 Diabetes to Improve Diabetes Care
Acronym: T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Ellis, Ph.D., Professor of Family Medicine and Public Health Sciences Wayne State University School of Medicine, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 066115B3E; R01DK059067 (NIH)
Record Dates: First submitted 2016-04-28; First posted 2016-05-03 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Type 1 Diabetes
Keywords: insulin dependent diabetes mellitus; adolescents and young adults; stress reduction; metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cognitive Behavioral Therapy; Mindfulness-Based Stress Reduction; Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive Behavioral Therapy (Experimental): Hains' adaptation of cognitive behavioral therapy for adolescents and young adults with type 1 diabetes
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Mindfulness Based Stress Reduction (Experimental): Sabinga's adaptation of Mindfulness Based Stress Reduction for adolescents and young adults with type 1 diabetes
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Diabetes Support and Education (Active Comparator): Investigator developed peer support group and diabetes education
  Interventions: Behavioral: Diabetes Support and Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will attend group therapy sessions, once a week for 9 weeks. The focus of these sessions will be the thought-emotion-behavior linkages as outlined by cognitive-behavioral theory. Activities will illustrate how thoughts affect emotions and behaviors, the application of these activities to current stressors, and strategies to apply these new skills to future stressors.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Mindfulness Based Stress Reduction — Participants will attend group therapy sessions, once a week for 9 weeks. The focus of these sessions will be understanding how to gain control over one's thoughts and feelings using relaxation, meditation, and other mindfulness-based techniques. Activities will focus on the instruction and practice of mindfulness techniques, such as meditation and yoga, and the application of these practices to everyday activities.
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction
Behavioral: Diabetes Support and Education — Participants will attend group therapy sessions, once a week for 9 weeks. Participants will receive diabetes education via a support group format. The focus of these sessions will be peer group social support and non-adherence diabetes education topics (e.g., emergency preparedness, smoking and diabetes).
  Other Names: DSE
  Arms: Diabetes Support and Education

SUMMARY:
Adolescence and young adulthood may be particularly stressful developmental periods due to the numerous transitions into new roles and the need for increased independence. Stress can affect metabolic control in older adolescents and young adults with T1D directly through its impact on cortisol and other hormones that affect insulin metabolism.

The proposed study is a pilot randomized clinical trial using a three-group randomized, repeated measures design to assess the efficacy of two treatments (Mindfulness Based Stress Reduction (MBSR) and Cognitive Behavioral Therapy or (CBT) versus an attention control condition for older adolescents and young adults with poorly controlled Type 1 diabetes. As a pilot study, the goal of the research is to test recruitment and retention procedures, finalize intervention measures, training, and fidelity protocols, and estimate effect sizes for a larger clinical trial.

DETAILED DESCRIPTION:
This study will use a randomized, repeated measures design. A sample of 125 participants will be recruited and consented from the Children's Hospital of Michigan and outpatient diabetes clinics affiliated with the Detroit Medical Center. 108 will be randomized to one of three treatment conditions (remaining participants are expected to consent but not enroll or fail to initiate treatment). These participants will be enrolled in 3 cohorts of 30-36 participants.

Measures will be administered at 3 home-based study visits to maximize participant convenience. The initial study visit (Visit 1) will be scheduled at the beginning of the study. Visit 2 will coincide with the end of treatment which is approximately 3 months after the initial study visit. Visit 3 is the 3-month follow up and will be scheduled about 6 months after the initial study visit. At each visit, participants will complete questionnaires assessing their current diabetes management, stressors, quality of life, mental health, and demographic characteristics. These questionnaires will be completed using Qualtrics accessed via the internet on a university laptop computer. A research assistant will download the participant's glucose meter to obtain the frequency of blood glucose testing during the two weeks preceding data collection. The research assistant will also assist participants with providing a blood sample via fingerstick (HbA1c) and saliva samples by mouth (cortisol, Visits 1 and 2 only). All participants will be asked to take part in an exit interview at Visit 3 to obtain feedback on the treatment they received.

After Visit 1, participants will be randomized using a 1:1:1 ratio to MBSR, CBT, or Diabetes Support and Education (DSE). All three treatments are group format meeting (10-12 participants per group) for nine consecutive weeks at a location convenient to the participants. In MBSR treatment focuses on the instruction and practice of mindfulness techniques, such as meditation and yoga, and the application of these practices to everyday activities. CBT utilizes activities to understand how thoughts affect emotions and behaviors, the application of these activities to current stressors, and strategies to apply these new skills to future stressors. The DSE group is the attention control condition; DSE participants will receive diabetes education via a support group format. All group sessions will be audiotaped for treatment fidelity monitoring and assessment. There are no planned research interventions for the DSE group.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 16 years, 0 months to 20 years, 11 months
2. Diagnosed with type 1 diabetes for at least six months
3. Poor metabolic control as defined by HbA1c >=9%

Exclusion Criteria:

1. Mental health conditions that might compromise data integrity (e.g., developmental delay, psychosis, suicidality)
2. Co-morbid medical condition resulting in atypical diabetes management (e.g., cystic fibrosis)
3. Inability to speak or read English

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Metabolic Control | Change from Baseline at 3 months, Change from Baseline at 6 months
  Hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Regimen Adherence (objective) | Change from Baseline at 3 months, Change from Baseline at 6 months
  Frequency of Glucose Meter Testing
Regimen Adherence (daily diary) | Change from Baseline at 3 months, Change from Baseline at 6 months
  24 Hour Recall of Diabetes Adherence Behavior
Regimen Adherence (self-reported) | Change from Baseline at 3 months, Change from Baseline at 6 months
  Diabetes Management Scale (DMS)
Psychological Stress (general) | Change from Baseline at 3 months, Change from Baseline at 6 months
  Perceived Stress Scale (PSS)
Psychological Stress (diabetes-related) | Change from Baseline at 3 months, Change from Baseline at 6 months
  Diabetes Stress Questionnaire (DSQ)
Psychological Stress (attitudes) | Change from Baseline at 3 months, Change from Baseline at 6 months
  Hassles and Uplifts Scale
Diabetes Quality of Life | Change from Baseline at 3 months, Change from Baseline at 6 months
  Diabetes Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Ellis, Ph.D, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University School of Medicine, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No